CLINICAL TRIAL: NCT00710268
Title: A Phase I, Open Label, Dual Centre Study To Assess The Safety And Tolerability Of AZD2281 In Combination With Bevacizumab (Avastin®) In Patients With Advanced Solid Tumours
Brief Title: Study to Assess Safety & Tolerability of AZD2281 in Combination With Bevacizumab in Patients With Advanced Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D0810C00022
Record Dates: First submitted 2008-06-30; First posted 2008-07-04 (Estimated); Last update posted 2015-01-14 (Estimated); Status verified 2015-01

CONDITIONS: Neoplasm Metastasis
Keywords: Bevacizumab; Poly(ADP ribose) polymerases; Metastatic Solid Tumours; PARP inhibitor
MeSH Terms: conditions — Neoplasm Metastasis | interventions — olaparib; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Dose Escalation Study 50, 100, 200, 400 mg
  Interventions: Drug: AZD2281; Drug: Bevacizumab

INTERVENTIONS:
Drug: AZD2281 — Oral Capsule, Dose Escalation 50, 100, 200, 400 mgContinuous twice daily dosing
  Other Names: Olaparib
Drug: Bevacizumab — IV administration10 mg/kg every 14 days
  Other Names: Avastin

SUMMARY:
Phase I, open label, dual centre, dose finding study to evaluate the safety and tolerability of continuous twice daily oral dosing with AZD2281 when administered in combination with Bevacizumab 10mg/kg given every 2 weeks to patients with advanced solid tumours.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed metastatic cancer, not amenable to surgery or radiation therapy with curative intent
* Adequate bone marrow, kidney and liver function in accordance with laboratory parameters set out in the protocol
* Estimated life expectancy of at least 12 weeks

Exclusion Criteria:

* Disorders that may put the patient at risk of bleeding, including gastrointestinal perforation, intra-abdominal abcess, major surgery of the chest or abdomen, previous haemorrhage, coughing up blood or thrombotic event
* Hypertension (high blood pressure) or significant cardiovascular disease
* Hypersensitivity to Chinese hamster ovary cell products or other recombinant or humanised antibodies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-06; Primary Completion 2009-03 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
safety and tolerability of twice daily oral doses of AZD2281 when administered in combination with Bevacizumab to patients with advanced solid tumours by assessment of adverse events, vital signs, ECG, clinical chem, haematology, urinalysis and phys exam | various timepoints.

SECONDARY OUTCOMES:
To compare exposure to AZD2281 when given alone and in combination with Bevacizumab, by assessment of appropriate derived PK parameters | various timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: James Carmichael, BSc MBChB MD FRCP, Study Director — KuDOS Pharmaceuticals Ltd; Malcolm Ranson, Principal Investigator — Christie Hospital, Manchester, UK
Locations (2):
- United Kingdom (2):
  - Research Site, Manchester
  - Research Site, Oxford

REFERENCES:
- See also: D0810C00022_CSR_Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1675&filename=D0810C00022.pdf